CLINICAL TRIAL: NCT05396742
Title: A Partially Randomized, Sequential Cohort, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Subcutaneous Ravulizumab Coadministered With rHuPH20 in Healthy Adult Volunteers
Brief Title: Pharmacokinetic Study of Ravulizumab Administered Subcutaneously With Recombinant Human Hyaluronidase PH20 (rHuPH20) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ALXN1210-HV-105; 2017-004931-35 (EudraCT Number)
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: ALXN1210; Pharmacokinetic; Pharmacodynamic; Safety; Immunogenicity; Ravulizumab; rHuPH20
MeSH Terms: interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Cohort 1 (Experimental): Participants received a single dose of ravulizumab SC 400 (milligrams) mg .
  Interventions: Drug: Ravulizumab
- Cohort 2 (Experimental): Participants received a single dose of ravulizumab SC 500 mg/rHuPH20 10000 units.
  Interventions: Drug: Ravulizumab; Drug: rHuPH20
- Cohort 3 (Experimental): Participants received a single dose of ravulizumab SC 1000 mg/rHuPH20 20000 units.
  Interventions: Drug: Ravulizumab; Drug: rHuPH20
- Cohort 4 (Experimental): Participants received a single dose of ravulizumab SC 2000 mg/rHuPH20 40000 units.
  Interventions: Drug: Ravulizumab; Drug: rHuPH20
- Cohort 5 (Experimental): Participants received a single dose of ravulizumab intravenously (IV) 400 mg.
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Ravulizumab — Solution for infusion or injection, as applicable
  Other Names: Ultomiris; ALXN1210
Drug: rHuPH20 — Solution for infusion
  Other Names: Recombinant human hyaluronidase PH20
  Arms: Cohort 2; Cohort 3; Cohort 4

SUMMARY:
The main objectives of this study were to estimate the absolute bioavailability of ravulizumab/rHuPH20 subcutaneous (SC) and to assess the safety and tolerability of ravulizumab/rHuPH20 SC.

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight between 60 and 90 kilogram (kg), inclusive, and body mass index within the range 18 through 29.9 kg/square meter, inclusive.
* Negative serum pregnancy test at screening and Day -1
* Male participants and females of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (at least 1 of which must be a barrier method) while on treatment and for up to 8 months after last dose of study drug.
* QT interval corrected using the Fridericia's formula (QTcF) ≤450 milliseconds (msec) for male participants and ≤470 msec for female participants at screening and prior to dosing on Day 1.
* Documented vaccination with meningococcal conjugate vaccine (MCV4) at least 56 days and not more than 2 years, 4 months prior to dosing.
* Vaccination with serogroup B meningococcal vaccine at least 56 days prior to dosing on Day 1, with a booster administered at least 28 days prior to dosing on Day 1, with at least 28 days between the first and second injections.

Key Exclusion Criteria:

* Current or recurrent disease (for example, cardiovascular, hematological, neurological, endocrine, immunological, rheumatological, renal, hepatic or gastrointestinal or other conditions) that or could affect clinical assessments or clinical laboratory evaluations.
* Current or relevant history of physical or psychiatric illness that are not stable or may require a change in treatment, use of prohibited therapies during the study or make the participant unlikely to fully comply with the requirements of the study or complete the study, or any condition that presents undue risk from the investigational product or study procedures.
* Any other significant disease or disorder which, in the opinion of the Investigator, may put the participant at risk.
* Documented history of allergy to penicillin or cephalosporin.
* History of significant allergic reaction (for example, anaphylaxis or angioedema) to any product (for example, food, pharmaceutical).
* Use of prescription medications (excluding oral contraceptives) within 14 days prior to dosing on Day 1, except with prior approval of the Sponsor.
* Regular use of nonprescription, over-the-counter medications, including herbal remedies and supplements, within 14 days prior to dosing on Day 1. Multivitamins, paracetamol (acetaminophen) ≤2 grams (g) per day, and topical skin products without significant systemic absorption are allowed.
* Positive urine drug toxicology screen at screening or on Day -1.
* Alcohol consumption within 48 hours prior to study drug administration or positive alcohol breath test on Day -1.
* Donation of plasma within 7 days prior to dosing on Day 1. Donation or loss (excluding volume drawn at screening) of more than 50 milliliters (mL) of blood within 30 days prior to dosing or more than 499 mL of blood within 56 days prior to dosing on Day 1.
* Female participants who are breastfeeding.
* Participants who are in intimate and prolonged contact with (defined as living under the same roof or providing personal care to) people younger than 2 years of age or older than 65 years of age, or who are either immunocompromised or have one of the following underlying medical conditions: anatomic or functional asplenia (including sickle cell disease); congenital complement, properdin, factor D, or primary antibody deficiencies; acquired complement deficiencies (for example, those receiving eculizumab); or human immunodeficiency virus (HIV).
* Participants who are one of the following:

  1. Professionals exposed to environments of greater risk for meningococcal disease
  2. Research, industrial, and clinical laboratory personnel who are routinely exposed to N meningitidis
  3. Military personnel during recruit training
  4. Daycare center workers
  5. Those living on a college or university campus
  6. Those who plan to travel during the course of the study to or have travelled to endemic areas for meningococcal meningitis (for example, India, Sub-Saharan Africa, pilgrimage to Saudi Arabia for Hajj) within 6 months prior to dosing
* Immunization with a live-attenuated vaccine 28 days prior to dosing on Day 1 or planned vaccination during the course of the study (except for the vaccination planned by the study protocol). Immunization with inactivated or recombinant influenza vaccine is permitted.
* Prior exposure to ravulizumab or eculizumab.
* Major surgery or hospitalization within 90 days prior to dosing on Day 1.
* History of allergy or hypersensitivity to excipients of ravulizumab (for example, polysorbate 80), rHuPH20, or other hyaluronidases.
* Currently smokes >10 cigarettes daily (former smokers may be permitted to enroll at the Investigator's discretion) and is unwilling to refrain from smoking while a resident in the clinical research unit or comply with the smoking restrictions.
* History of illicit drug abuse, history of significant alcohol abuse within 1 year prior to the screening visit, or clinical evidence of substance and/or alcohol abuse within the 2 years before screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants who met all inclusion and no exclusion criteria were assigned unique numbers for enrollment and randomization. Randomization was only used when cohorts were enrolled in parallel.
Pre-assignment Details: A total of 108 potential participants were screened (including 5 rescreened and 59 rejects [screen fail]). A total of 49 participants were ultimately treated in this study.
Groups:
- Cohort 1: Participants received a single dose of ravulizumab 400 mg (milligrams) subcutaneously.
- Cohort 2: Participants received a single dose of ravulizumab 500 mg/recombinant human hyaluronidase PH20 (rHuPH20) 10000 units subcutaneously.
- Cohort 3: Participants received a single dose of ravulizumab 1000 mg/rHuPH20 20000 units subcutaneously.
- Cohort 4: Participants received a single dose of ravulizumab 2000 mg/rHuPH20 40000 units subcutaneously.
- Cohort 5: Participants received a single dose of ravulizumab 400 mg intravenously.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 7 | 12 | 12 | 12 | 6
Received at Least 1 Dose of Study Drug | 7 | 12 | 12 | 12 | 6
Completed | 7 | 12 | 12 | 12 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who receive at least 1 dose of study drug.
Groups:
- Cohort 1: Participants received a single dose of ravulizumab 400 mg subcutaneously.
- Cohort 2: Participants received a single dose of ravulizumab 500 mg/rHuPH20 10000 units subcutaneously.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 7 | 12 | 12 | 12 | 6 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (7.41) | 27.5 (5.11) | 28.9 (6.99) | 29.5 (7.57) | 28.8 (4.75) | 28.8 (6.34)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0 | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0 | 0 | 0 | 0
  Adults (18-64 years) | 7 | 12 | 12 | 12 | 6 | 49
  From 65-84 years | 0 | 0 | 0 | 0 | 0 | 0
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 7 | 3 | 0 | 16
  Male | 5 | 8 | 5 | 9 | 6 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 12 | 12 | 11 | 6 | 47
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 1 | 2 | 0 | 1 | 4
  Black or African American | 2 | 1 | 0 | 0 | 1 | 4
  White | 4 | 9 | 9 | 11 | 3 | 36
  Other | 1 | 1 | 1 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Absolute Bioavailability Of Ravulizumab Subcutaneous (SC)/rHuPH20
Description: Dose-normalized area under the serum concentration versus time curve from 0 extrapolated to infinity (AUC0-inf) and body weight-adjusted AUC0-inf for the ravulizumab/rHuPH20 SC cohorts were compared with the 400 mg ravulizumab intravenous (IV) cohort to determine absolute bioavailability. Geometric mean ratios of the AUC0-inf parameter were calculated for each group. Absolute bioavailability is reported as the geometric mean ratio, which was defined as the ratio of geometric means for the dose-normalized AUC0-inf parameter (with and without body-weight adjustment) for the ravulizumab SC cohort divided by that for the ravulizumab IV cohort.
Time Frame: Day 1 (after first dose) to Day 200
Population: The Pharmacokinetics (PK) Population included all participants who had sufficient serum concentration data to enable the calculation of PK parameters of at least area under the serum concentration versus time curve (AUC). For this outcome measure, the Number of Participants Analyzed includes the participants from both the IV group and the respective SC group.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent bioavailability
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 12 | 18 | 18 | 18
Percent bioavailability
  Dose-normalized AUC0-inf | 64 [44 to 92] | 73 [57 to 94] | 77 [57 to 102] | 84 [63 to 113]
  Body weight-adjusted and dose-normalized AUC0-inf | 63 [46 to 85] | 69 [57 to 84] | 70 [55 to 90] | 81 [63 to 104]

2. Primary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was reported as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. Serious AEs (SAEs) were defined as any untoward medical occurrence that, at any dose resulted in death, life threatening, required hospitalization, resulted in persistent disability or incapacity, resulted in birth defect, or other situations. A summary of serious and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Day 1 (after first dose) up to Day 200 (including safety follow up)
Population: The Safety Population included all participants who receive at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 7 | 12 | 12 | 12 | 6
Participants
  TEAEs | 7 | 11 | 12 | 10 | 5
  SAEs | 0 | 0 | 0 | 0 | 0
  Discontinuations due to TEAEs | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Relative Bioavailability Of Ravulizumab SC/rHuPH20 Compared With Ravulizumab SC
Description: Dose-normalized AUC0-inf and body weight-adjusted AUC0-inf for the ravulizumab/rHuPH20 SC cohorts were compared with the 400 mg ravulizumab SC cohort to determine relative bioavailability. Geometric mean ratios of the AUC0-inf parameter were calculated for each group. Relative bioavailability is reported as the geometric mean ratio, which was defined as the ratio of the geometric means for the dose-normalized AUC0-inf parameter (with and without body-weight adjustment) for the ravulizumab/rHuPH SC cohort divided by that for the ravulizumab SC cohort.
Time Frame: Day 1 (after first dose) to Day 200
Population: The PK Population included all participants who had sufficient serum concentration data to enable the calculation of PK parameters of at least AUC. For this outcome measure, the Number of Participants Analyzed includes the participants from both the ravulizumab/rHuPH SC cohort and the respective ravulizumab SC cohort.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent bioavailability
Arm/Group | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 18 | 18 | 18
Percent bioavailability
  Dose-normalized AUC0-inf | 115 [91 to 145] | 120 [91 to 158] | 132 [100 to 175]
  Body weight-adjusted and dose-normalized AUC0-inf | 109 [90 to 134] | 112 [88 to 142] | 129 [101 to 165]

4. Secondary Outcome: Maximum Percent Change From Baseline (PCFB) In Serum Levels Of Total Complement Component 5 (C5) Concentrations
Description: The highest (maximum difference) mean (standard deviation [SD]) PCFB at up to Day 200 is reported. Baseline was defined as the last available value prior to the first drug administration. Change from Baseline was calculated as observed value minus the baseline value. PCFB was calculated as change from baseline divided by baseline multiplied by 100.
Time Frame: Baseline, Up to Day 200
Population: The Pharmacodynamics (PD) Population included all participants who had sufficient free C5 concentration data that enabled the evaluation of the PD effects.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 12 | 12 | 12 | 6
Percent change | 92.12 (58.332) | 98.68 (27.659) | 107.46 (45.769) | 133.48 (35.782) | 112.90 (27.878)

5. Secondary Outcome: Maximum PCFB In Serum Levels Of Free C5 Concentrations
Description: The highest (maximum difference) mean (SD) PCFB at up to Day 200 is reported. Baseline was defined as the last available value prior to the first drug administration. Change from Baseline was calculated as observed value minus the baseline value. PCFB was calculated as change from baseline divided by baseline multiplied by 100.
Time Frame: Baseline, Day 200
Population: The PD Population included all participants who had sufficient free C5 concentration data that enabled the evaluation of the PD effects.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 12 | 12 | 12 | 6
Percent Change | -96.83 (4.783) | -99.48 (0.349) | -99.84 (0.116) | -99.90 (0.00) | -99.90 (0.00)

6. Secondary Outcome: Maximum PCFB In Ex Vivo Chicken Red Blood Cell (cRBC) Hemolysis Activity
Description: as for outcome 5
Time Frame: Baseline, Up to Day 200
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 12 | 12 | 12 | 6
Percent change | -58.07 (19.382) | -77.68 (23.765) | -80.74 (28.153) | -99.35 (0.684) | -98.52 (1.790)

ADVERSE EVENTS:
Time Frame: Day 1 (after first dose) up to Day 200 (including safety follow up)
Description: The Safety Population included all participants who receive at least 1 dose of study drug.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/12 | 0/12 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/12 | 0/12 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 7/7 | 11/12 | 12/12 | 10/12 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1 (N=7) | Cohort 2 (N=12) | Cohort 3 (N=12) | Cohort 4 (N=12) | Cohort 5 (N=6)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (4) | 1 (1)
Injection site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 6 (11) | 4 (4) | 4 (4) | 3 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1/2 (1) | 0/4 (0) | 0/7 (0) | 1/3 (1) | 0/0 (0) — The N for this adverse event has been adjusted to the number of females in the study as it is a sex-specific event.
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 2 (4)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Medical device site reaction (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hangover (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 1 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 3 (3) | 6 (6) | 4 (4) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1/2 (1) | 0/4 (0) | 0/7 (0) | 0/3 (0) | 0/0 (0) — The N for this adverse event has been adjusted to the number of females in the study as it is a sex-specific event.
Laryngitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infections (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular access site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal cyst (Reproductive system and breast disorders) | 0/2 (0) | 0/4 (0) | 1/7 (1) | 0/3 (0) | 0/0 (0) — The N for this adverse event has been adjusted to the number of females in the study as it is a sex-specific event.
Vaginal discharge (Reproductive system and breast disorders) | 0/2 (0) | 1/4 (1) | 0/7 (0) | 0/3 (0) | 0/0 (0) — The N for this adverse event has been adjusted to the number of females in the study as it is a sex-specific event.
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menstruation normal (Investigations) | 0/2 (0) | 0/4 (0) | 1/7 (1) | 0/3 (0) | 0/0 (0) — The N for this adverse event has been adjusted to the number of females in the study as it is a sex-specific event.
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT05396742/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT05396742/SAP_001.pdf